CLINICAL TRIAL: NCT03321045
Title: PET Imaging With 89Zr-Trastuzumab for Prediction of HER2 Targeted Therapy Effectiveness
Brief Title: Positron Emission Tomography (PET) Imaging With Zirconium-89 (89Zr)-Trastuzumab for Prediction of HER2 Targeted Therapy Effectiveness
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Suzanne E. Lapi, PhD, Associate Professor of Radiology and Director, Cyclotron Facility, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-170220004; UAB (Other: UAB Department of Radiology)
Record Dates: First submitted 2017-10-19; First posted 2017-10-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: 89Zr-Trastuzumab, HER2 Imaging
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [89Zr]-Df-Trastuzumab (Experimental): [89Zr]-Df-Trastuzumab [89Zr]-Df-Trastuzumab will be administered intravenously. The administered dose will be 2 millicurie (mCi) at the time of injection. The amount of injected drug is 5 mg of Trastuzumab. 5-6 days post injection the patients will undergo PET/MRI imaging.
  Interventions: Drug: [89Zr]-Df-Trastuzumab; Diagnostic Test: PET/MRI Imaging

INTERVENTIONS:
Drug: [89Zr]-Df-Trastuzumab — [89Zr]-Df-Trastuzumab will be administered intravenously. The administered dose will be 2 mCi at the time of injection. The amount of injected drug is 5 mg of Trastuzumab.
Diagnostic Test: PET/MRI Imaging — 5-6 days post injection the patients will undergo PET/MRI imaging.

SUMMARY:
Our goal is to investigate the use of 89Zr-trastuzumab as a HER2 imaging agent to determine which patients are likely to respond to targeted HER2 agents as single agent therapy. We are proposing to perform a pilot study with goals of demonstrating the feasibility of imaging breast cancer patients with 89Zr-trastuzumab-PET/MRI, evaluating the relationship between tumor 89Zr-trastuzumab uptake and in vitro positivity of HER2, assessing the relationship between 89Zr-trastuzumab uptake and response to HER2 therapy.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age.
* Diagnosis of HER2 positive breast cancer as defined by to American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) 2018 guidelines: Immunohistochemistry (IHC) 3+ OR Single prove In situ hybridization (ISH) with average HER2 copy number >= 6 OR dual probe ISH with both average HER2 copy number >= 4 AND HER2 to CEP17 ratio >=2
* Patients eligible for radiation therapy or systemic therapy using a regimen containing at least one anti-HER2 agent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 and 1
* Ejection fraction greater than 50% by echocardiogram or multiple-gated acquisition (MUGA) scans

Exclusion Criteria:

* Inability to provide informed consent
* Pregnancy
* Inability to lie still for the imaging study
* Weight over 350 lbs., due to the scanner bore size
* Contraindication for MRI study (e.g. non-removable metal implants or certain tattoos)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Estimated)
Dates: Start 2017-11-21 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Investigate the use of [89Zr]-Df-Trastuzumab as a HER2 imaging agent | 24 months
  To measure the diagnostic quality (with standardized uptake values) of PET/MRI imaging with [89Zr]-Df-Trastuzumab in patients with newly diagnosed breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne E Lapi, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- The Kirklin Clinic, Birmingham, Alabama, United States